CLINICAL TRIAL: NCT00655057
Title: SPECT Brain Imaging as a Bio-Marker of Major Depression
Brief Title: Effects of Antidepressant Therapy on Brain Dopamine Transporter Activity in People With Major Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R34MH070753 (NIH); R34MH070753 (NIH); DATR A3-NSS
Record Dates: First submitted 2008-04-07; First posted 2008-04-09 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Depression
Keywords: Dopamine Transporter; Biomarker; SPECT Brain Imaging; Antidepressant Therapy
MeSH Terms: conditions — Depression | interventions — Dexetimide; Cognitive Behavioral Therapy; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Healthy participants will undergo TRODAT-1 SPECT imaging.
  Interventions: Procedure: TRODAT-1 single photon emission computed tomographic (SPECT) imaging
- 2 (Experimental): Participants with depression will undergo TRODAT-1 SPECT imaging and treatment with s-citalopram.
  Interventions: Drug: S-citalopram; Procedure: TRODAT-1 single photon emission computed tomographic (SPECT) imaging
- 3 (Active Comparator): Participants with depression will undergo TRODAT-1 SPECT imaging and treatment with cognitive behavioral therapy.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Procedure: TRODAT-1 single photon emission computed tomographic (SPECT) imaging

INTERVENTIONS:
Drug: S-citalopram — Participants will take 10 to 30 mg of s-citalopram daily for 12 weeks.
  Arms: 2
Behavioral: Cognitive behavioral therapy (CBT) — Participants will attend twice weekly CBT sessions for 2 weeks and then once weekly sessions for 10 weeks. Sessions will focus on modifying thoughts and behaviors that may contribute to depression.
  Arms: 3
Procedure: TRODAT-1 single photon emission computed tomographic (SPECT) imaging — Participants' striatal dopamine transporter (DAT) levels will be measured using [99mTc]TRODAT-1 SPECT with magnetic resonance imaging (MRI) co-localization on two separate occasions. Participants with depression will undergo TRODAT-1 SPECT imaging immediately before and after 12 weeks of their assigned treatment. Healthy participants will undergo TRODAT-1 SPECT imaging at baseline and 12 weeks later.

SUMMARY:
This study will examine changes in brain dopamine transporter activity before and after antidepressant therapy.

DETAILED DESCRIPTION:
Depression is a serious psychiatric disorder that affects about 10% of the adult population in the United States in a given year. Common symptoms of depression include a persistent down mood and disinterest in previously enjoyed activities, often causing strain on work, social, and family life. A person's depression can be attributed to a variety of causes, including physiological and sociological factors. Among physiological factors, dopamine (DA), a chemical associated with feelings of happiness and pleasure, may play a key role in the onset of depression and may also be involved in the beneficial effect of antidepressant medication. Recent studies have found that people with depression have increased DA transporter (DAT) levels in a specific region of the inner brain called the striatum. The increased DAT levels might reflect alterations in central DA function. Treatment for depression with selective serotonin reuptake inhibitor (SSRI) antidepressant therapy may help in returning DAT levels to normal and in improving depressive symptoms. Using single photon emission computed tomography (SPECT) imaging, this study will examine changes in brain DAT activity in people with depression before and after they receive SSRI antidepressant therapy or cognitive behavioral therapy (CBT).

Participation in this study will last about 14 weeks and will involve participants who are healthy and depressed. All participants will first undergo baseline assessments that will include a medical history, questions about current and past health, a physical exam, a blood draw, a urine sampling, and an electrocardiogram (ECG). After completing the baseline assessments, participants will undergo a TRODAT-1 SPECT scan, which will involve an injection of TRODAT-1 (a radioactive agent to measure DA) and, after a 3-hour break, a 75-minute SPECT scan. If necessary, participants may also be asked to have a magnetic resonance imaging (MRI) brain scan after completing the SPECT scan.

Participants with depression will then be assigned randomly to undergo 12 weeks of treatment with either the antidepressant medication s-citalopram or CBT. Participants assigned to take s-citalopram will return for study visits weekly for 2 weeks, every other week for 6 weeks, and then monthly for 4 weeks. During study visits, participants will receive their medication, answer questions about depression and medication side effects, and occasionally fill out general health questionnaires. Participants receiving CBT will attend twice weekly sessions for 2 weeks and then once weekly sessions for 10 weeks. Sessions will focus on modifying thoughts and behaviors that may contribute to depression. After 12 weeks, all participants will be re-evaluated by a study doctor and, if still in good health, will undergo a repeat TRODAT-1 SPECT scan.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of major depressive episode (MDE) or major depressive disorder (MDD)
* Drug free of psychotropic medication for more than 6 months before study entry
* 17-item Hamilton Depression Scale (HAM-D17) score of greater than 16
* Woman of childbearing age with a negative pregnancy test within 48 hours of study entry
* Absence of DSM-IV Axis I diagnosis as determined by Structured Clinical Interview for DSM Disorders (SCID)

Exclusion Criteria:

* DSM-IV Axis I diagnosis other than MDE
* History of mania
* Current alcohol or drug abuse, or alcohol or drug dependence within 6 months before study entry
* History of sensitivity or intolerance to s-citalopram
* Medical contraindication to the use of s-citalopram
* Unstable medical condition (e.g., angina pectoris, untreated hypertension)
* Pregnant or breastfeeding
* Woman of childbearing potential not using a medically acceptable form of birth control
* Actively suicidal or requiring hospitalization
* Requiring additional psychotropic drug therapy
* History of transient ischemic attacks
* History of cerebral infarction (including lacunar infarct with symptoms that last more than 24 hours)
* History of Binswanger's disease (or a history of hypertensive encephalopathy)
* History of intracranial hemorrhage
* History of head trauma with loss of consciousness
* History of encephalitis
* History of extended exposure to known neurotoxin (e.g., cyanide, carbon monoxide)
* Uncontrolled metabolic disorder (e.g., thyroid disease, diabetes mellitus)
* History of cognitive impairment other than MDE
* History of normal pressure hydrocephalus
* History of cancer metastatic to the central nervous system
* History of Parkinson's disease or other basal ganglia disease
* History of Guillain-Barre syndrome (chronic or relapsing polyneuropathy)
* Inability to undergo an MRI scan
* History of DSM-IV Axis I Mood Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2005-10; Primary Completion 2009-08 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jay D. Amsterdam, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Depression Research Unit - University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Groups:
- Healthy Participants: Healthy participants will undergo TRODAT-1 SPECT imaging.
  TRODAT-1 single photon emission computed tomographic (SPECT) imaging: Participants' striatal dopamine transporter (DAT) levels will be measured using [99mTc]TRODAT-1 SPECT with magnetic resonance imaging (MRI) co-localization on two separate occasions. Participants with depression will undergo TRODAT-1 SPECT imaging immediately before and after 12 weeks of their assigned treatment. Healthy participants will undergo TRODAT-1 SPECT imaging at baseline and 12 weeks later.
- Patients With Depression Without CBT: Participants with depression will undergo TRODAT-1 SPECT imaging and treatment with s-citalopram.
  S-citalopram: Participants will take 10 to 30 mg of s-citalopram daily for 12 weeks.
  TRODAT-1 single photon emission computed tomographic (SPECT) imaging: Participants' striatal dopamine transporter (DAT) levels will be measured using [99mTc]TRODAT-1 SPECT with magnetic resonance imaging (MRI) co-localization on two separate occasions. Participants with depression will undergo TRODAT-1 SPECT imaging immediately before and after 12 weeks of their assigned treatment. Healthy participants will undergo TRODAT-1 SPECT imaging at baseline and 12 weeks later.
- Patients With Depression: CBT and SPECT: Participants with depression will undergo TRODAT-1 SPECT imaging and treatment with cognitive behavioral therapy.
  Cognitive behavioral therapy (CBT): Participants will attend twice weekly CBT sessions for 2 weeks and then once weekly sessions for 10 weeks. Sessions will focus on modifying thoughts and behaviors that may contribute to depression.
  TRODAT-1 single photon emission computed tomographic (SPECT) imaging: Participants' striatal dopamine transporter (DAT) levels will be measured using [99mTc]TRODAT-1 SPECT with magnetic resonance imaging (MRI) co-localization on two separate occasions. Participants with depression will undergo TRODAT-1 SPECT imaging immediately before and after 12 weeks of their assigned treatment. Healthy participants will undergo TRODAT-1 SPECT imaging at baseline and 12 weeks later.
Period: Overall Study
Arm/Group | Healthy Participants | Patients With Depression Without CBT | Patients With Depression: CBT and SPECT
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Participants | Patients With Depression Without CBT | Patients With Depression: CBT and SPECT | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Customized [unit: participants]
Sex/Gender, Customized [unit: participants]
Race and Ethnicity Not Collected — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Change in Dopamine Transporter Binding
Time Frame: Measured at Weeks 0 and 12
Population: as for baseline characteristics
Arm/Group | Healthy Participants | Patients With Depression Without CBT | Patients With Depression: CBT and SPECT
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 Years
Description: The investigator has succumb to serious health issues which prevents him from physically inputting data in the system. The study team is no longer at the university and despite all efforts to contact them in order to enter data on the investigator's behalf, data are not available.
Arm/Group | Healthy Participants | Patients With Depression Without CBT | Patients With Depression: CBT and SPECT
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Data is unavailable for the following reasons: Principal Investigator has succumb to serious health issues preventing data input, and study team is no longer with the university and is unreachable to input data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes